CLINICAL TRIAL: NCT00538811
Title: Interferon-gamma With Interferon Alpha and Ribavirin for Hepatitis C Patients Who Are Non-responders to Interferon Alpha Plus Ribavirin
Brief Title: Interferon-gamma With Interferon Alpha and Ribavirin for Hepatitis C Non-responders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 648-Med
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Hepatitis C; Genotype 3; Non-responders; Relapsers
MeSH Terms: conditions — Hepatitis C | interventions — Introns; Ribavirin; Interferon-gamma; Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Interferon alpha, ribavirin, interferon gamma
  Interventions: Drug: interferon alpha-2b, ribavirin, interferon-gamma,
- 2 (Active Comparator): Interferon alpha, ribavirin, amantadine
  Interventions: Drug: interferon alpha-2b, ribavirin, amantadine

INTERVENTIONS:
Drug: interferon alpha-2b, ribavirin, interferon-gamma,
  Arms: 1
Drug: interferon alpha-2b, ribavirin, amantadine
  Arms: 2

SUMMARY:
When administered simultaneously, interferon-alpha 2b + interferon-gamma result in dramatic antiviral synergy.Ribavirin has shown to enhance interferon-gamma levels in patients with chronic hepatitis C treated with interferon-alpha. Enhancement of immune responses, especially those related to type-1 T helper cell activity, may contribute to better efficacy in combining ribavirin with IFN-alpha for treatment of chronic hepatitis C. The aim of the present study is to evaluate the efficacy and safety of a triple regimen, a combination treatment with Interferon gamma, Interferon alfa-2b plus Ribavirin in patients who have not previously responded to interferon alpha in combination of ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Non-responders and relapsers to previous interferon and ribavirin therapy given for six months
* HCV genotype 3
* Compensated liver disease
* Hb ≥10 g/dl (females),≥11 g/dl (males)
* Platelets count ≥ 100,000 / cubic mm
* Neutrophils count ≥1,500/cubic mm
* ≥18 years to ≤ 70 years.
* At least one abnormal ALT value in the last year.
* TSH level within normal limits.
* Non pregnant adult females.
* Absence of drug or alcohol abuse.
* Informed consent given by the patient

Exclusion Criteria:

* Patient younger than 18 yrs and older than 70 yrs.
* Hepatitis B or HIV co-infection.
* Severe renal dysfunction or creatinine clearance less than 50 ml/min
* Pregnant women or breast feeding women.
* Suspected hypersensitivity to Interferon alpha, gamma or ribavirin.
* Decompensated liver cirrhosis.
* History or any other evidence of other causes of CLD other than hepatitis C infection ( like hemochromatosis,, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposure, Wilson's disease,Drug induced liver disease)
* Active malignant disease.
* Any known pre-existing medical condition that could interfere with subject's participation or completion of study such as psychiatric condition, seizures disorder requiring medications, co existing heart diseases, lung diseases, poorly controlled diabetes, auto immune diseases, gout)
* History of interferon and/or ribavirin intolerance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zaigham Abbas, FCPS, FACG, Principal Investigator — The Aga Khan University Hospital
Locations (2):
- Pakistan (2):
  - Medicare Clinic, Karachi
  - The Aga Khan University Hospital, Karachi

REFERENCES:
- [Derived] Abbas Z, Raza S, Hamid S, Jafri W. Randomized controlled trial of interferon gamma versus amantadine in combination with interferon alpha and ribavirin for hepatitis C genotype 3 non-responders and relapsers. J Pak Med Assoc. 2012 Apr;62(4):338-43. PMID 22755276